CLINICAL TRIAL: NCT06754150
Title: Shoulder Innovations Clinical Data Registry
Acronym: SICDR
Status: Recruiting | Type: Observational
Sponsor: Shoulder Innovations (Industry)
Responsible Party: Sponsor
Other Study IDs: SICDR 31.0.1.1.1
Record Dates: First submitted 2024-12-13; First posted 2024-12-31 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Shoulder Arthroplasty
Keywords: Shoulder Arthroplasty; Shoulder Replacement; Anatomic Shoulder Arthroplasty; Reverse Shoulder Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this multi-center observational study is to collect long-term clinical outcome information for anatomic and reverse total shoulder arthroplasty (shoulder replacement).

DETAILED DESCRIPTION:
The study is a non-randomized, multi-center prospective registry that will collect standard-of-care data for patients who plan to receive or have received shoulder arthroplasty (anatomic or reverse) with a Shoulder Innovations (SI) Total Shoulder System device and consent to participate in the study. The study will evaluate short and long term clinical and radiographic outcomes associated with real-world use of the arthroplasty system from the implant procedure through 10 years post-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Plan to receive or has received a shoulder arthroplasty surgical procedure, with a minimum of one implanted Shoulder Innovations (SI) device component and be willing and able to complete post-operative visits as long as at least one SI device component remains implanted.
3. Able to provide informed consent prior to enrollment in the study (unless a waiver has been obtained).
4. Agree to and be able to consistently answer the specified Patient Reported Outcome Measures (PROM) pre-operatively and at each of the post-operative visits without the use of a translator.
5. Willing and able to comply with the requirements of the study protocol

Exclusion Criteria:

1. Participation in a clinical trial of an investigational drug or device that would confound the results of this trial. Participation in another observational registry is allowed provided there are no conflicting requirements to this trial.
2. Incarceration.
3. Any conditions, co-morbidities, restrictions, or obligations that would prohibit them from complying with the requirements of this study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (at least 18 years of age) of any gender undergoing a shoulder arthroplasty for any diagnosis/condition with at least one SI Total Shoulder System component enrolled at participating sites
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2039-12 (Estimated); Study Completion 2039-12 (Estimated)

PRIMARY OUTCOMES:
Durability of the device component implant | From the implant procedure until 10 years post-operatively
  Assessment of the SI device component will be made at specified intervals using x-rays to check how long the device component can stay implanted with or without a revision surgery.

SECONDARY OUTCOMES:
Change in range of motion (ROM) post-operatively at specified timepoints as compared to baseline | From baseline (pre-operatively) until 10 years post-operatively
Change in ASES score post-operatively at specified timepoints as compared to baseline | From baseline (pre-operatively) until 10 years post-operatively
  Patients will complete the ASES questionnaire (American Shoulder and Elbow Surgeons Shoulder Score) to evaluate pain and activities of daily living.
Change in SANE score post-operatively at specified timepoints as compared to baseline | From baseline (pre-operatively) until 10 years post-operatively
  Patients will complete the SANE questionnaire (Single Assessment Numeric Evaluation) to rate their affected shoulder as a percentage of normal.
Change in PROMIS Global-10 score post-operatively at specified timepoints as compared to baseline | From baseline (per-operatively) until 10 years post-operatively
  Patients will complete the PROMIS Global-10 questionnaire (Patient-Reported Outcome Measurement Information System Global-10) to evaluate pain and activities of daily living.
Evaluation of radiographic images for radiolucent lines, implant stability and loosening | From baseline (pre-operatively) until 10 years post-operatively
Rate of intra-operative and post-operative adverse device effects (ADEs)/complications | From the implant procedure until 10 years post-operatively

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - St. Vincent's Orthopedics, Birmingham, Alabama
  - California Pacific Orthopaedics, San Francisco, California
  - Western Orthopaedics, Denver, Colorado
  - Connolly Orthopedics, Bradenton, Florida
  - Georgia Bone and Joint, Newnan, Georgia
  - North Shore Physicians Group, Peabody, Massachusetts